CLINICAL TRIAL: NCT00498836
Title: A Multicentre, Dose Finding, Phase II Study of CP-4055 in Combination With Sorafenib in Patients With Metastatic Malignant Melanoma
Brief Title: Multicentre, Dose Finding, Ph II,CP-4055 in Comb. With Sorafenib - Patients With Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clavis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP4055-203
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-08

CONDITIONS: Malignant Melanoma
Keywords: CP-4055; Elacyt; Cancer; Metastatic; Malignant melanoma; Combination treatment; Sorafenib; Nexavar
MeSH Terms: conditions — Melanoma; Neoplasms; Neoplasm Metastasis | interventions — 5'-oleoyl cytarabine; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CP-4055 — CP-4055 5mg/mL for infusion, dose: 200 mg/m2/day, schedule d1-5 q4w, 30 minutes IV infusion
  Other Names: ELACYT (TM)
Drug: Sorafenib (Nexavar) — Sorafenib 200 mg tablets, dose: 400 mg/day, daily dosing
  Other Names: Nexavar

SUMMARY:
Patients with metastatic malignant melanoma will receive CP-4055 200 mg/m2/day intravenously (IV) on Day 1-5 every four weeks and sorafenib 400 mg b.i.d. (twice daily) every day until complete response or disease worsening/progressing.

DETAILED DESCRIPTION:
This is a multicentre clinical study conducted in the USA and in Europe. It is an open label study designed to investigate objective tumor response, the time to progression (TTP) and the duration of tumor response in patients with metastatic malignant melanoma when treated with CP-4055 in combination with sorafenib (Nexavar®). The safety and tolerability of the treatment will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological or cytological confirmed stage IV or unresectable stage III non-ocular malignant melanoma who have or have not undergone prior chemotherapy for the treatment of melanoma
2. Measurable disease according to Response Criteria In Solid Tumors (RECIST)
3. Performance Status 0 - 1 according to ECOG (Eastern Cooperative Oncology Group) Performance Status
4. Age 18 years or more
5. Life expectancy > 3 months
6. Signed informed consent
7. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must have a negative serum or urine pregnancy test within 2 weeks prior to beginning treatment on this study
8. Male and female patients must use acceptable contraceptive methods for the duration of time on study, and males also for 3 months after the last CP-4055 dose
9. Adequate haematological and biological functions

Exclusion Criteria:

1. Known brain metastases
2. Diagnosis of ocular malignant melanoma
3. Radiotherapy to more than 30 % of bone marrow
4. Participation in another therapeutic clinical study within 30 days of enrolment or during this clinical study
5. Requirement of concomitant treatment with a non-permitted medication:

   * Alternative drugs
   * High doses of vitamins
6. History of allergic reactions to ara-C or egg
7. History of allergic reactions attributed to compounds of similar chemical or biological composition to sorafenib
8. Presence of any serious concomitant systemic disorders incompatible with the clinical study (e.g. uncontrolled inter-current illness including ongoing or active infection)
9. Presence of any significant central nervous system or psychiatric disorder(s) that would hamper the patient's compliance
10. Pregnancy, breastfeeding or absence of adequate contraception for both male and female fertile patients
11. Known positive status for HIV and/or hepatitis B or C
12. Drug and/or alcohol abuse
13. Any reason why, in the investigator's opinion, the patient should not participate
14. Prior treatment with CP-4055 and/or sorafenib
15. Significant history of cardiac disease, including any of the following:

    * Uncontrolled hypertension
    * Unstable angina pectoris
    * Congestive heart failure
    * Myocardial infarction within the past 6 months
    * Unstable ventricular arrhythmia
    * Other cardiac arrhythmia
16. Condition that impairs ability to swallow pills
17. Tendency of bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
• Objective tumour response | October 2008

SECONDARY OUTCOMES:
• Time to progression | October 2008
• Duration of tumour response | October 2008
• Safety and tolerability of treatment | October 2008

CONTACTS AND LOCATIONS:
Overall Officials: Svein Dueland, MD, Principal Investigator — The Norwegian Radium Hospital, Oslo, Norway
Locations (6):
- United States (2):
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Cancer Therapy and Research Center, Institute for Drug Development, San Antonio, Texas
- The Norwegian Radium Hospital, Oslo, Norway
- Sweden (3):
  - Lund University Hospital, Lund
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala